CLINICAL TRIAL: NCT04840563
Title: Evaluation of Surface Refractive Index Shift and Lens Absorption / Adsorption of Tear Components of Commercially Available Kalifilcon A Lenses Compared to Dailies Total1 and Precision1
Brief Title: Surface Refractive Index Shift and Lens Absorption/Adsorption of Tear Components of Kalifilcon A Lenses vs Dailies Total1 and Precision1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROC2-21-007
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Habitual Soft Contact Lens Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Kalifilcon A lenses (Experimental): Commercially available kalifilcon A lenses (Bausch + Lomb)
  Interventions: Device: Kalifon A
- Dailies Total1 (Active Comparator): Dailies Total1 (Alcon)
  Interventions: Device: Dailies Total1
- Precision1 (Active Comparator): Precision1 (Alcon)
  Interventions: Device: Precision1

INTERVENTIONS:
Device: Kalifon A — Commercially available kalifilcon A lenses
  Arms: Kalifilcon A lenses
Device: Dailies Total1 — Dailies Total1
  Arms: Dailies Total1
Device: Precision1 — Precision1
  Arms: Precision1

SUMMARY:
Approximately 10 habitual soft contact lens wearing participants will be enrolled in this bilateral, randomized, double-masked (participant and investigator masked) repeated measures insertion study. All participants will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If participants satisfy all eligibility criteria and none of the exclusion criteria, participants will insert study lenses in random, successive order according to unique randomization schedules that will be provided to each Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older and have full legal capacity to volunteer.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Surface refractive index shifts | 10 minutes
  Immediately following lens removal, the right eye worn lenses for each subject will be measured for surface refractive index on the refractometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch Site 001, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided